CLINICAL TRIAL: NCT00006604
Title: Phase I/II, Open-Label, Pharmacokinetic and Safety Study of a Novel Protease Inhibitor (BMS 232632, Atazanavir, ATV, Reyataz) in Combination Regimens in Antiretroviral Therapy (ART)-Naive and -Experienced HIV-Infected Infants, Children, and Adolescents
Brief Title: Atazanavir Used in Combination With Other Anti-HIV Drugs in HIV-Infected Infants, Children, and Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1020A; 10037 (Registry Identifier: DAIDS ES); IMPAACT P1020A; PACTG P1020-A; ACTG P1020-A
Record Dates: First submitted 2000-12-06; First posted 2001-08-31 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2016-03

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Drug Therapy, Combination; Drug Administration Schedule; HIV Protease Inhibitors; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Pharmacokinetics; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Step I: Group 1 (Experimental): Group 1 enrolled participants between 91 days of age and 2 years of age. They received ATV (powder) and two NRTIs.
  ATV Dose Tested: 310 mg/m^2, 620 mg/m^2; Final Dose: Not Established
  Interventions: Drug: ATV
- Step I: Group 2 (Experimental): Group 2 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (powder) and two NRTIs.
  ATV Dose Tested: 310 mg/m^2, 620 mg/m^2; Final Dose: Not Established
  Interventions: Drug: ATV
- Step I: Group 3 (Experimental): Group 3 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (capsule) and two NRTIs.
  ATV Dose Tested: 310 mg/m^2, 415 mg/m2, 520 mg/m^2; Final Dose: 520 mg/m^2
  Interventions: Drug: ATV
- Step I: Group 4 (Experimental): Group 4 enrolled participants between 13 years and 1 day of age and 21 years of age. They received ATV (capsule) and two NRTIs.
  ATV Dose Tested: 310 mg/m^2, 520 mg/m^2, 620 mg/m^2; Final Dose: 620 mg/m^2
  Interventions: Drug: ATV
- Step I: Group 5 (Experimental): Group 5 enrolled participants between 91 days of age and 2 years of age. They received ATV (powder), ritonavir, and two NRTIs.
  ATV Dose Tested: 310 mg/m^2; Final Dose: 310 mg/m^2
  Interventions: Drug: ATV; Drug: Ritonavir
- Step I: Group 5a (Experimental): Group 5a enrolled participants between 91 days of age and 180 days of age. They received ATV (powder), ritonavir, and two NRTIs.
  ATV Dose Tested: 310 mg/m^2; Final Dose: 310 mg/m^2
  Interventions: Drug: ATV; Drug: Ritonavir
- Step I: Group 6 (Experimental): Group 6 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (powder), ritonavir, and two NRTIs.
  ATV Dose Tested: 310 mg/m^2; Final Dose: 310 mg/m^2
  Interventions: Drug: ATV; Drug: Ritonavir
- Step I: Group 7 (Experimental): Group 7 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (capsule), ritonavir, and two NRTIs.
  ATV Dose Tested: 310 mg/m^2, 205 mg/m^2; Final Dose: 205 mg/m^2
  Interventions: Drug: ATV; Drug: Ritonavir
- Step I: Group 8 (Experimental): Group 8 enrolled participants between 13 years and 1 day of age and 21 years of age. They received ATV (capsule), ritonavir, and two NRTIs.
  ATV Dose Tested: 310 mg/m^2, 205 mg/m^2; Final Dose: 205 mg/m^2
  Interventions: Drug: ATV; Drug: Ritonavir

INTERVENTIONS:
Drug: ATV — Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
Drug: Ritonavir — Administered as 100 mg capsules or oral solution.
  Arms: Step I: Group 5; Step I: Group 5a; Step I: Group 6; Step I: Group 7; Step I: Group 8

SUMMARY:
The purpose of this study was to find a safe and tolerable dose of the protease inhibitor (PI) atazanavir (ATV), with or without a low-dose boost of the PI ritonavir (RTV), when taken with other anti-HIV drugs in HIV infected infants, children, and adolescents.

Advancements in anti-HIV drugs for HIV infected children and adolescents have been hard to make, in part because these patients often do not take the drugs as prescribed. ATV may be a better option because it is available in the form of powder which children and adolescents may be more willing to take regularly. Using a low dose of RTV as a boosting agent for ATV may also increase the chances of virologic response of highly active antiretroviral treatment (HAART)-experienced patients. This study aimed to find safe and tolerable doses of ATV with or without low-dose RTV boost in infants, children, and adolescents. For this study, participants were enrolled in the United States and South Africa.

DETAILED DESCRIPTION:
Advancements in HAART for HIV-infected children and adolescents are hindered by patient nonadherence. The availability of a powder formulation and the once-daily dosing schedule make ATV an attractive agent for improved adherence in pediatric treatment regimens. This study was designed to provide pharmacokinetic (PK) data to guide dosing recommendations for ATV, when given concurrently with or without low-dose RTV boost, in infants, children, and adolescents. During the study, the safety and tolerance of ATV (with or without low-dose RTV) were closely monitored, and virologic efficacy data were obtained.

There were two parts to this study. Step I took place in the United States and South Africa, and were further divided into two sets of groups, Parts A and B. Part A participants received ATV only and Part B participants received ATV with low-dose RTV boost. All participants received ATV once a day with 2 other antiretroviral drugs (not provided by the study). In Part B only, participants received ATV with a low dose of RTV. Participants were placed into 1 of 8 groups (Groups 1 to 4 for Part A; Groups 5 to 8 for Part B) with respect to age and study drug formulation. Participants in Groups 1 and 5 were infants between ages 3 months and 1 day (91 days) and 2 years (less than or exactly 730 days) and took ATV in powder form. Participants in Groups 2, 3, 6, and 7 were children between 2 years and 1 day (731 days) old and 13 years old. Groups 2 and 6 received ATV in powder form, while Groups 3 and 7 received the capsule form. Patients in Groups 4 and 8 were adolescents between 13 years and 1 day old and 21 years old (not including the 22nd birthday) and took ATV in capsule form. As of 01/02/2008 a new group, 5A was opened for enrollment. Participants in Group 5A were between 3 months and 6 months old and took ATV in powder form plus a low-dose RTV booster.

For each group, enrollment started with five participants per group. All participants were evaluated for PK and safety criteria, adjusting the dose of ATV until one was found that passes both sets of criteria. Then five additional participants were enrolled, with enrollment continuing for each group once all participants within that group meet the PK criteria. For groups receiving RTV (Groups 5 to 8), additional criteria must be met for each dose of ATV studied. In addition to the PK and safety evaluations, 24-hour post-dose concentrations (Cmin) were monitored in the first 10 participants enrolled for a dose of ATV before more participants were enrolled and studied at that same dose. Note that in Protocol Version 5.0, South African (S.A.) sites were allowed to enroll patients in study groups 3,4,5,6,7,8. As a result, the study design has been modified to further stratify study groups 3, 4, 5, 6, 7, 8 (at the final recommended dose), by country, i.e., U.S.A. versus S.A., such that 10 evaluable study subjects will be accrued in parallel to each study group-country cohort.

Clinic visits will be every 4 weeks through Week 48, then every 8 weeks until the last participant to enroll in the study has reached Week 96 of his/her treatment. If, after 56 weeks, a participant has a toxic reaction to a nucleoside/tide reverse transcriptase inhibitor (NRTI) in their medication regimen, the regimen may be changed to a different NRTI. At every visit, participants will undergo a complete medical history and physical exam, cardiac conduction evaluation, and urine and blood collection. Participants of childbearing age will have a pregnancy test performed at each visit.

Step II will only be open to South African subjects who are virologically responding to treatment when the last enrollee into either part of Step I (Part A or Part B) has completed 96 weeks of treatment (end of Step I) . All such participants will be given ATV in capsule form at the same dose they received at the end of Step I, as well as the other antiretrovirals they were receiving during Step I. Step II will continue until ATV is approved in South Africa and readily available by individual prescription, and participants will have a study visit every 12 weeks.

Note that the following ATV doses were independently evaluated for each group during the dose-finding stage based on the description above: Group 1 ATV Powder (310mg/m^2, 620mg/m^2); Group 2 ATV Powder (310mg/m^2, 620mg/m^2); Group 3 ATV Capsule (310mg/m^2, 415mg/m^2, 520mg/m^2); Group 4 ATV Capsule (310mg/m^2, 520mg/m^2, 620mg/m^2); Group 5 ATV Powder + RTV (310mg/m^2); Group 6 ATV Powder +RTV (310mg/m^2); Group 7 ATV Capsule + RTV (310mg/m^2, 205mg/m^2); Group 8 ATV Capsule + RTV (310mg/m^2, 205mg/m^2); Group 5A ATV Powder + RTV (310mg/m^2). All these dosing groups are presented in Participant Flow groups to show the total number of participants enrolled, but only the participants enrolled at the final group doses are presented in the subsequent results.

The following groups satisfied the safety and PK guidelines specified in the protocol: Groups 3,4,6,7,8. Groups 5 and 5A did not satisfy the protocol-defined pharmacokinetic criteria. There was considerable inter-subject variability in systemic exposures in this age group, such that a dose escalation to 415mg/m^2 may have resulted in ATV exposures greater than 90,000 ng*hr/mL in some children. Thus, a further dose increase in Groups 5 and 5A was not attempted.

These are the final dose for each group: Groups 1 and 2 (Final dose was not established); Group 3 ATV Capsule (520mg/m^2); Group 4 ATV Capsule (620mg/m^2); Group 5 ATV Powder (310mg/m^2) + RTV; Group 6 ATV Powder (310mg/m^2) +RTV; Group 7 ATV Capsule (205mg/m^2) + RTV; Group 8 ATV Capsule (205mg/m^2) + RTV; Group 5A ATV Powder (310mg/m^2) + RTV.

ELIGIBILITY:
Inclusion Criteria for Step I:

* Age: 91 days to 21 years of age (not including the 22nd birthday).
* A confirmed diagnosis of HIV infection defined by the current definition of the IMPAACT Virology Core Laboratory Committee. More information about this criterion can be found in the protocol.
* Viral load greater than or equal to 5,000 copies/mL
* Any CDC clinical classification and immune status
* Antiretroviral treatment-naïve or -experienced study candidates must be able to add two new NRTIs as part of their new therapy in this protocol, or have genotypic evidence of sensitivity to two NRTIs (the NRTIs must be used in combinations recommended in the Guidelines for the Use of Antiretroviral Agents in Pediatric and Adolescent HIV Infection). More information about this criterion can be found in the protocol.
* Study candidates must show evidence of retained phenotypic sensitivity to ATV (resistance index ratio of less than 10) when the subject has failed (after at least 12 weeks of therapy) two or more courses of PI containing regimens. More information about this criterion can be found in the protocol.
* Demonstrated ability and willingness to swallow study medications
* Study candidate, parent, or legal guardian must be able and willing to provide signed informed consent
* Female participants who are sexually active and able to become pregnant must use two methods of birth control. More information about this criterion can be found in the protocol.
* Males participating in the study must not attempt to impregnate a female, or participate in sperm donation programs. Males engaging in sexual activity that could lead to pregnancy must use a condom.
* Study candidates with a history of undefined syncope will require a complete cardiac conduction evaluation at screening [e.g., ECG, 24-hour monitoring (Holter), and exercise test (if age appropriate)]. This evaluation must rule-out any cardiac conduction abnormalities.

Exclusion Criteria for Step I:

* Active hepatitis
* Presence of an acute serious/invasive infection requiring therapy at the time of enrollment
* Hypersensitivity to any component of the formulation of ATV
* Chemotherapy for active malignancy
* Pregnant or breastfeeding
* Any clinically significant diseases (other than HIV infection) or clinically significant findings during the screening medical history or physical examination that, in the clinician's opinion, would compromise the outcome of this study
* Any laboratory or clinical toxicity greater than Grade 2 at entry
* Documented history of cardiac conduction abnormalities or significant cardiac dysfunction
* History of undefined syncope that cannot be ruled out as related to cardiac conduction abnormalities
* Family history of prolonged QTc-interval syndrome, Brugada syndrome, or right-ventricular (RV) dysplasia
* Corrected QTc-Interval greater than 440 msec at screening
* Prolonged PR-Interval greater than 0.200 seconds (200 ms) on ECG at screening (study candidates greater than or equal to 13 years of age)
* PR-Interval greater than 98th percentile on ECG at screening (study candidates less than 13 years of age)
* Cardiac rhythm abnormalities:

  1. A type I second-degree atrioventricular (AV) block (Mobitz type I heart-block) occurring during waking hours on ECG at screening
  2. A type II second-degree AV-block (Mobitz type II heart-block) at any time on ECG at screening
  3. A complete AV-block at any time on ECG at screening
  4. A heart rate less than the 2nd percentile for age of the normal heart rate range on ECG at screening
* Prolonged therapy with intravenous pentamidine for acute Pneumocystis Carinii Pneumonia (PCP) within three months of entry

Inclusion Criteria for Step II:

* Any South African subject enrolled into either part of Step I, who is virologically successful by Week 96 of when the last study participant enrolled into the respective part of Step I
* Female participants who are sexually active and able to become pregnant must continue using two methods of birth control. More information about this criterion can be found in the protocol.
* Males who continue participation in the study must not attempt to impregnate a woman, or participate in sperm donation programs. Males engaging in sexual activity that could lead to pregnancy must use a condom.

Exclusion Criteria for Step II:

* A South African participant who meets any of the criteria for treatment discontinuation by Week 96 of when the last participant enrolled into either part of Step I
* A South African participant who meets any of the exclusion criteria from Step I by Week 96 of when the last participant enrolled into either part of Step I

Ages: 91 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 195 (Actual)
Dates: Start 2000-11; Primary Completion 2011-10 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Rutstein, MD, Study Chair — Children's Hospital of Philadelphia
Locations (36):
- United States (32):
  - UAB Pediatric Infectious Diseases CRS, Birmingham, Alabama
  - Usc La Nichd Crs, Alhambra, California
  - University of California, UC San Diego CRS, La Jolla, California
  - Miller Children's Hosp. Long Beach CA NICHD CRS, Long Beach, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Univ. of California San Francisco NICHD CRS, San Francisco, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Columbus Regional HealthCare System, The Med. Ctr., Columbus, Georgia
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Tulane Univ. New Orleans NICHD CRS, New Orleans, Louisiana
  - Univ. of Maryland Baltimore NICHD CRS, Baltimore, Maryland
  - Johns Hopkins Univ. Baltimore NICHD CRS, Baltimore, Maryland
  - Boston Medical Center Ped. HIV Program NICHD CRS, Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey
  - Nyu Ny Nichd Crs, New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Bronx-Lebanon Hospital Center NICHD CRS, The Bronx, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - Philadelphia IMPAACT Unit CRS, Philadelphia, Pennsylvania
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
  - Children's Med. Ctr. Dallas, Dallas, Texas
  - Texas Children's Hospital CRS, Houston, Texas
  - Children's Hosp. of the King's Daughters, Infectious Disease, Norfolk, Virginia
  - Childrens Hosp. of the Kings Daughters, Norfolk, Virginia
  - Seattle Children's Research Institute CRS, Seattle, Washington
- Puerto Rico (2):
  - Univ. Hosp. Ramón Ruiz Arnau, Dept. of Peds., Bayamón
  - San Juan City Hosp. PR NICHD CRS, San Juan
- South Africa (2):
  - Soweto IMPAACT CRS, Johannesburg, Gauteng
  - Shandukani CRS, Johannesburg, Gauteng

REFERENCES:
- [Background] Rutstein RM, Samson P, Fenton T, Fletcher CV, Kiser JJ, Mofenson LM, Smith E, Graham B, Mathew M, Aldrovani G; PACTG 1020A Study Team. Long-term safety and efficacy of atazanavir-based therapy in HIV-infected infants, children and adolescents: the Pediatric AIDS Clinical Trials Group Protocol 1020A. Pediatr Infect Dis J. 2015 Feb;34(2):162-7. doi: 10.1097/INF.0000000000000538. PMID 25232777
- [Background] Kiser JJ, Rutstein RM, Samson P, Graham B, Aldrovandi G, Mofenson LM, Smith E, Schnittman S, Fenton T, Brundage RC, Fletcher CV. Atazanavir and atazanavir/ritonavir pharmacokinetics in HIV-infected infants, children, and adolescents. AIDS. 2011 Jul 31;25(12):1489-96. doi: 10.1097/QAD.0b013e328348fc41. PMID 21610486
- [Background] Aldrovandi G, Samson P, Fenton T, Schnittman S, Rutstein R, Ortiz A and the Pediatric AIDS Clinical Trial 1020A Group. Resistance to Atazanavir (ATV), Lopinavir (LPV), Tenofovir (TFV) Among Heavily Experienced Pediatric Patients. 12th International Symposium on HIV and Emerging Infectious Diseases in Toulon, France, June 2002.
- [Background] Aldrovandi G, Samson P, Fenton T, Schnittman S, and Rutstein R for the P1020A Team. Genotypic and phenotypic resistance to BMS232632 (Atazanavir-ATV), among heavily experienced pediatric patients who were ATV-naïve. 9th Conference on Retroviruses and Opportunistic Infections, February 24 - 28, 2002, Seattle, WA.
- [Background] Kiser J, Rutstein R, Aldrovandi G, Samson P, Graham B, Schnittman S, Smith M, Mofenson L, Fletcher C, and the PACTG 1020A Study Team. Pharmacokinetics of atazanavir/ritonavir in HIV-infected infants, children, and adolescents: PACTG 1020A. 12th Conference on Retroviruses and Opportunistic Infections, Boston, MA, February 2005.
- [Background] Kiser J, Rutstein R, Samson P, Graham B, Aldrovandi G, Mofenson L, Smith E, Zhang J, Biguenet S, Fletcher C, and the P1020A team. Atazanavir dosing conversion and pharmacokinetics in HIV-infected children switching from atazanavir powder to capsules. 12 th International Workshop on Clinical Pharmacology of HIV Therapy, Miami, Florida, April 2011.
- [Background] Meyers T, Rutstein R, Samson P, Violari A, Palmer M, Kiser J, Fletcher C, Fenton T, Mofenson L, Graham B, Schnittman S, Horga M, Aldrovandi G, for the PACTG 1020A Study. Treatment responses to atazanavir-containing HAART in a drug-naïve pediatric population in South Africa. 15th Conference on Retroviruses and Opportunistic Infections, Boston, MA, February 2008.
- [Background] Rutstein R, Samson P, Aldrovandi G, Graham B, Schnittman S, Fletcher C, Kiser J, Smith E, Mofenson L, Fenton T, and the PACTG 1020A Study Team. Effect of atazanavir on serum cholesterol and triglyceride levels in HIV-infected infants, children, and adolescents: PACTG 1020A. 12th Conference on Retroviruses and Opportunistic Infections, Boston, MA, February 2005.
- [Background] Rutstein R, Samson P, Fenton T, Kiser J, Fletcher C, Schnittman S, Mofenson L, Smith E, Graham B, Aldrovandi G, PACTG 1020A Study. The NIH PACTG Protocol 1020A: ATAZANAVIR (ATV), +/- RITONAVIR in HIV-Infected Infants, Children and Adolescents. Presented at the 14th Conference on Retrovirus and Opportunistic Infection (CROI), Los Angeles, CA, February, 2007.
- [Background] Samson P, Rutstein R, Schnittman S, Ortiz A, Graham B, Fenton T, Aldrovandi G and the Pediatric AIDS Clinical Trials Group P1020A Study Team. Effects of Antiretroviral (ARV) Exposure and Genotypic (Geno) Mutations in Predicting Phenotypic Resistance (PRS) to Atazanavir (ATV), Lopinavir (LPV), and Tenofovir (TDF) in Patients Naïve to these Drugs. 13th International Symposium on HIV and Emerging Infectious Diseases, Toulon, France, June 2004.
- [Background] Samson P, Rutstein R, Fenton T, Kiser J, Fletcher C, Schnittman S, Mofenson L, Smith E, Graham B, Aldrovandi G, and the PACTG 1020A Study Team. Changes in cholesterol and triglyceride levels among pediatric subjects treated with atazanavir, with or without ritonavir boosting: the 1020A NIH PACTG protocol. 13th Conference on Retroviruses and Opportunistic Infections, Denver, CO, February 2006.
- See also: DAIDS Toxicity Table for Grading Severity of Pediatric (> 3 mos of age) Adverse Experiences April, 1994. — http://rsc.tech-res.com/Document/safetyandpharmacovigilance/Table_for_Grading_Severity_of_Pediatric_AEs_Over3MonthsAge_v03.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of First Enrollment: 16 November 2000; Date of Last Enrollment: 22 December 2009
Groups:
- Group 1: ATV Dose: Powder (310mg/m^2); Group 1: ATV Dose: Powder (620mg/m^2): Group 1 enrolled participants between 91 days of age and 2 years of age. They received ATV (powder) and two NRTIs.
- Group 2: ATV Powder (310mg/m^2); Group 2: ATV Powder (620mg/m^2): Group 2 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (powder) and two NRTIs.
- Group 3: ATV Capsule (310mg/m^2): Group 3 enrolled participants between 2 years and 1 day of age and 13 years of age. They will received ATV (capsule) and two NRTIs.
- Group 3: ATV Capsule (415mg/m^2): Group 3 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (capsule) and two NRTIs.
- Group 3: ATV Capsule (520mg/m^2): Group 3 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (capsule) and two NRTIs.
  Note: This is the final recommended dose for this group.
- Group 4: ATV Capsule (310mg/m^2); Group 4: ATV Capsule (520mg/m^2): Group 4 enrolled participants between 13 years and 1 day of age and 21 years of age. They received ATV (capsule) and two NRTIs.
- Group 4: ATV Capsule (620mg/m^2): Group 4 enrolled participants between 13 years and 1 day of age and 21 years of age. They received ATV (capsule) and two NRTIs.
  Note: This is the final recommended dose for this group.
- Group 5: ATV Powder (310mg/m^2) + RTV: Group 5 enrolled participants between 91 days of age and 2 years of age. They received ATV (powder), ritonavir, and two NRTIs.
  Note: This is the final recommended dose for this group.
- Group 5a: ATV Powder (310mg/m^2) + RTV: Group 5a enrolled participants between 91 days of age and 180 days of age. They received ATV (powder), ritonavir, and two NRTIs.
  Note: This is the final recommended dose for this group.
- Group 6: ATV Powder (310mg/m^2) + RTV: Group 6 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (powder), ritonavir, and two NRTIs.
  Note: This is the final recommended dose for this group.
- Group 7: ATV Capsule (310mg/m^2) + RTV: Group 7 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (capsule), ritonavir, and two NRTIs.
- Group 7: ATV Capsule (205mg/m^2) + RTV: Group 7 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (capsule), ritonavir, and two NRTIs.
  Note: This is the final recommended dose for this group.
- Group 8: ATV Capsule (310mg/m^2) + RTV: Group 8 enrolled participants between 13 years and 1 day of age and 21 years of age. They received ATV (capsule), ritonavir, and two NRTIs.
- Group 8: ATV Capsule (205mg/m^2) + RTV: Group 8 enrolled participants between 13 years and 1 day of age and 21 years of age. They received ATV (capsule), ritonavir, and two NRTIs.
  Note: This is the final recommended dose for this group.
Period: Overall Study
Arm/Group | Group 1: ATV Dose: Powder (310mg/m^2) | Group 1: ATV Dose: Powder (620mg/m^2) | Group 2: ATV Powder (310mg/m^2) | Group 2: ATV Powder (620mg/m^2) | Group 3: ATV Capsule (310mg/m^2) | Group 3: ATV Capsule (415mg/m^2) | Group 3: ATV Capsule (520mg/m^2) | Group 4: ATV Capsule (310mg/m^2) | Group 4: ATV Capsule (520mg/m^2) | Group 4: ATV Capsule (620mg/m^2) | Group 5: ATV Powder (310mg/m^2) + RTV | Group 5a: ATV Powder (310mg/m^2) + RTV | Group 6: ATV Powder (310mg/m^2) + RTV | Group 7: ATV Capsule (310mg/m^2) + RTV | Group 7: ATV Capsule (205mg/m^2) + RTV | Group 8: ATV Capsule (310mg/m^2) + RTV | Group 8: ATV Capsule (205mg/m^2) + RTV
Started | 6 | 2 | 5 | 6 | 5 | 5 | 21 | 5 | 5 | 25 | 21 | 12 | 26 | 6 | 24 | 6 | 15
Completed | 4 | 2 | 1 | 1 | 3 | 2 | 12 | 2 | 4 | 6 | 13 | 6 | 22 | 0 | 14 | 1 | 6
Not Completed | 2 | 0 | 4 | 5 | 2 | 3 | 9 | 3 | 1 | 19 | 8 | 6 | 4 | 6 | 10 | 5 | 9
Not completed — Met study objective - no further FU | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Randomization entry error-no RX, no FU | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Severe debilitation, unable to continue | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 5 | 0 | 2 | 1 | 0 | 2 | 0 | 0
Not completed — Subj/Parent not able to get to clinic | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 3 | 0 | 0
Not completed — Site closing | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 0 | 1 | 2 | 2 | 0 | 1 | 3 | 2 | 0 | 1 | 2 | 1 | 0 | 1
Not completed — Subj/parent not willing to adhere to req | 0 | 0 | 1 | 3 | 0 | 0 | 3 | 1 | 0 | 6 | 3 | 0 | 0 | 2 | 3 | 3 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Other Reason | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants accrued and treated at the dose ultimately selected for their groups.
  NOTE: (1) Final Dose not established for Grps 1, 2; (2) Grp 5a started with n=12, but (1) participant inadvertently enrolled,never received ATV, final n=11; (3) Grp 8 started with n=15, but (1) participant inadvertently enrolled, never received ATV, final n=14.
Groups:
- Step I: Group 3 (ATV Final Dose: 520mg/m^2 Capsule): Group 3 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (capsule) and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  ATV Final Recommended Dose: 520mg/m^2
- Step I: Group 4 (ATV Final Dose: 620mg/m^2 Capsule): Group 4 enrolled participants between 13 years and 1 day of age and 21 years of age. They received ATV (capsule) and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  ATV Final Recommended Dose: 620mg/m^2
- Step I: Group 5 (ATV Final Dose: 310mg/m^2 Powder + RTV): Group 5 enrolled participants between 91 days of age and 2 years of age. They received ATV (powder), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended Dose: 310mg/m^2
- Step I: Group 5a (ATV Final Dose: 310mg/m^2 Powder + RTV): Group 5a enrolled participants between 91 days of age and 180 days of age. They received ATV (powder), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended Dose: 310mg/m^2
- Step I: Group 6 (ATV Final Dose: 310mg/m^2 Powder + RTV): Group 6 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (powder), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended Dose: 310mg/m^2
- Step I: Group 7 (ATV Final Dose: 205mg/m^2 Capsule + RTV): Group 7 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (capsule), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended Dose: 205mg/m^2
- Step I: Group 8 (ATV Final Dose: 205mg/m^2 Capsule + RTV): Group 8 enrolled participants between 13 years and 1 day of age and 21 years of age. They received ATV (capsule), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended Dose: 205mg/m^2
- Total: Total of all reporting groups
Arm/Group | Step I: Group 3 (ATV Final Dose: 520mg/m^2 Capsule) | Step I: Group 4 (ATV Final Dose: 620mg/m^2 Capsule) | Step I: Group 5 (ATV Final Dose: 310mg/m^2 Powder + RTV) | Step I: Group 5a (ATV Final Dose: 310mg/m^2 Powder + RTV) | Step I: Group 6 (ATV Final Dose: 310mg/m^2 Powder + RTV) | Step I: Group 7 (ATV Final Dose: 205mg/m^2 Capsule + RTV) | Step I: Group 8 (ATV Final Dose: 205mg/m^2 Capsule + RTV) | Total
Number analyzed (Participants) | 21 | 25 | 21 | 11 | 26 | 24 | 14 | 142
Age, Continuous [Median (Full Range); unit: years] | 8.6 [6.3 to 12.5] | 14.3 [13.1 to 20.2] | 1.2 [0.3 to 2.0] | 0.4 [0.3 to 0.5] | 4.4 [2.0 to 12.0] | 9 [5.6 to 12.7] | 17 [13.9 to 21] | 7 [0.3 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 18 | 8 | 6 | 12 | 11 | 9 | 75
  Male | 10 | 7 | 13 | 5 | 14 | 13 | 5 | 67
Race/Ethnicity, Customized [Number; unit: participants]
  White Non-Hispanic | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 5
  Black Non-Hispanic | 14 | 17 | 18 | 10 | 18 | 17 | 8 | 102
  Hisp-Regardless of Race | 3 | 7 | 2 | 1 | 7 | 5 | 5 | 30
  More than one race | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3
  Unavailable | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
CD4 Count [Median (Full Range); unit: cells/mm^3] | 374 [105 to 963] | 286 [11 to 476] | 1306 [392 to 4875] | 2125 [583 to 2715] | 466 [62 to 1537] | 540 [24 to 1800] | 334 [1 to 548] | 457 [1 to 4875]
CD4 Percent [Median (Full Range); unit: percentage of total lymphocytes] | 18 [7 to 36] | 14 [1 to 39] | 19 [7 to 53] | 35 [10 to 46] | 16 [2 to 34] | 21 [1 to 43] | 19 [0 to 40] | 18 [0 to 53]
HIV-RNA [Median (Full Range); unit: log10 copies/ml] | 4.4 [3.5 to 5] | 4.7 [3.6 to 6.5] | 5 [4.4 to 5.6] | 5 [5 to 6.5] | 4.8 [4.1 to 5.1] | 4.5 [3.4 to 5] | 4.3 [3.5 to 5] | 4.8 [3.4 to 6.5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Safety Endpoint of Interest Attributed to ATV
Description: Total Bilirubin >= 5.1xULN, ECG Events and Other Grade 3+ toxicities attributed to study treatment.
  The AEs were graded by the clinicians according to the Division of AIDS (DAIDS) Toxicity Table (see references in the Protocol Section) as follows: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Potentially Life-Threatening, Grade 5=Death. Relationship to study treatment was determined by the study team.
Time Frame: From study entry up to week 96
Population: Patients accrued at the final recommended dose for each group.
Measure: Number; unit: participants
Groups:
- Step I: Group 3: ATV Dose: 520mg/m^2 Capsule: Group 3 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (capsule) and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  ATV Final Recommended Dose: 520mg/m^2
- Step I: Group 4: ATV Dose: 620mg/m^2 Capsule: Group 4 enrolled participants between 13 years and 1 day of age and 21 years of age. They received ATV (capsule) and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  ATV Final Recommended Dose: 620mg/m^2
- Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV: Group 5 enrolled participants between 91 days of age and 2 years of age. They received ATV (powder), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended Dose: 310mg/m^2
- Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV: Group 5a enrolled participants between 91 days of age and 180 days of age. They received ATV (powder), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended: 310mg/m^2
- Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV: Group 6 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (powder), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended Dose: 310mg/m^2
- Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV: Group 7 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (capsule), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended Dose: 205mg/m^2
- Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV: Group 8 enrolled participants between 13 years and 1 day of age and 21 years of age. They received ATV (capsule), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended Dose: 205mg/m^2
Arm/Group | Step I: Group 3: ATV Dose: 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 21 | 25 | 21 | 11 | 26 | 24 | 14
participants
  Total Bilirubin >= 5.1xULN | 1 | 4 | 0 | 0 | 0 | 4 | 4
  Increase in PR Interval-Grade 1 | 11 | 4 | 3 | 1 | 4 | 5 | 1
  Increase in PR Interval-Grade 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Heart Rate-Grade 2 | 2 | 1 | 3 | 1 | 1 | 4 | 0
  Heart Rate-Grade 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Increase in QTc Interval-Grade 3 | 1 | 0 | 0 | 1 | 1 | 0 | 0
  Other Grade 3+ Toxicities | 0 | 3 | 0 | 2 | 0 | 1 | 0

2. Primary Outcome: Number of Participants Who Died
Time Frame: From study entry up to week 96
Population: Participants accrued at the final recommended dose for each group.
Measure: Number; unit: participants
Groups:
- Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV: Group 5a enrolled participants between 91 days of age and 180 days of age. They received ATV (powder), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended Dose: 310mg/m^2
Arm/Group | Step I: Group 3: ATV Dose: 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 21 | 25 | 21 | 11 | 26 | 24 | 14
participants
  Death not attributed to ATV | 0 | 1 | 1 | 1 | 0 | 0 | 0
  Death attributed to ATV | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With HIV RNA <400 Copies/mL at Week 24
Description: Over the duration of the protocol, the assay used to determine Plasma HIV RNA levels was transitioned from the Amplicor HIV-1 Assay to the Amplicor HIV-1 Monitor 1.5 UltraSensitive Assay (Roche Molecular Systems, Branchburg, NJ) to finally the Abbott Real time HIV-1 RNA assay. The assays were performed according to the manufacturer's instructions in a laboratory accredited by the College of American Pathologists and certified by the NIH Virology Quality Assurance (VQA) in the United States, and VQA certified in South Africa.
Time Frame: Week 24
Population: Participants accrued at the final recommended dose for each group (with evaluable HIV-RNA data).
  Virologic response, defined as achieving HIV-RNA < 400 copies/mL and remaining on treatment, was analyzed using an 'intent-to-treat' (ITT) approach, in which children who discontinued study treatment for any reason were considered failures.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Step I: Group 6 : ATV Dose: 310mg/m^2 Powder + RTV: Group 6 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (powder), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended Dose: 310mg/m^2
- Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV: Group 7 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (capsule), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended: 205mg/m^2
Arm/Group | Step I: Group 3: ATV Dose: 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6 : ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 21 | 25 | 21 | 9 | 26 | 24 | 13
percentage of participants | 67 [43 to 85] | 44 [24 to 65] | 57 [34 to 78] | 44 [14 to 79] | 85 [65 to 96] | 67 [45 to 84] | 38 [14 to 79]

4. Secondary Outcome: Percentage of Participants With HIV RNA <400 Copies/mL at Week 48
Description: as for outcome 3
Time Frame: Week 48
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Step I: Group 3: ATV Dose: 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 21 | 25 | 21 | 11 | 26 | 24 | 14
percentage of participants | 62 [38 to 82] | 32 [15 to 54] | 71 [48 to 89] | 55 [23 to 83] | 85 [65 to 96] | 63 [41 to 81] | 29 [8 to 58]

5. Secondary Outcome: Percentage of Participants With HIV RNA <400 Copies/mL at Week 96
Description: as for outcome 3
Time Frame: Week 96
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Step I: Group 3: ATV Dose: 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 21 | 25 | 20 | 5 | 26 | 24 | 14
percentage of participants | 48 [26 to 70] | 20 [7 to 41] | 75 [51 to 91] | 20 [1 to 72] | 73 [52 to 88] | 63 [41 to 81] | 14 [2 to 43]

6. Primary Outcome: Pharmacokinetic (PK) Parameter: Area Under the Curve (AUC24h)
Description: Pharmacokinetics were determined by non-compartmental analysis and AUC0-24hr calculated by the linear trapezoidal method.
Time Frame: Week 1 (Day 7) Intensive PK-24hr (Pre-Dose, 1, 2, 3, 4, 6, 8, and 12 hours post-dose and the following day at 24-hours post-dose)
Population: Participants with intensive pharmacokinetic (PK) results at the final recommended dose for each group.
Measure: Median (Inter-Quartile Range); unit: ng*hr/mL
Groups:
- Step I: Group 5: ATV 310mg/m^2 Powder + RTV: Group 5 enrolled participants between 91 days of age and 2 years of age. They received ATV (powder), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended Dose: 310mg/m^2
Arm/Group | Step I: Group 3: ATV Dose: 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 20 | 21 | 17 | 11 | 21 | 21 | 14
ng*hr/mL | 40653 [25498 to 49784] | 51781 [43287 to 78946] | 44243 [27504 to 69168] | 38928 [12005 to 54783] | 52199 [39847 to 76995] | 45680 [35379 to 55407] | 42835 [37753 to 56663]

7. Primary Outcome: Pharmacokinetic (PK) Parameter: Minimum Plasma Concentration (C24)
Description: Pharmacokinetics were determined by non-compartmental analysis. C24 determined visually, except in the instance when the patient re-dosed the study medication prior to the 24 hour blood draw or the 24 hour level was not obtained, in which case the C24 was calculated from the elimination rate (ke) and the last measured concentration.
Time Frame: as for outcome 6
Population: Participants with intensive pharmacokinetic (PK) results at the final recommended dose for each group.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Step I: Group 3: ATV Dose: 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 20 | 21 | 17 | 11 | 21 | 21 | 14
ng/mL | 173 [99 to 317] | 510 [245 to 761] | 482 [194 to 627] | 596 [138 to 810] | 947 [521 to 1280] | 575 [389 to 858] | 885 [692 to 1491]

8. Primary Outcome: Pharmacokinetic (PK) Parameter: Maximum Plasma Concentration (Cmax)
Description: Pharmacokinetics were determined by non-compartmental analysis and Maximum concentration (Cmax) was determined visually.
Time Frame: Week 1 (Day 7) Intensive PK-24 hr (Pre-dose, 1, 2, 3, 4, 6, 8, and 12 hours post-dose and the following day at 24-hours post-dose)
Population: Participants with intensive pharmacokinetic (PK) results at the final recommended dose for each group.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- Step I: Group 3: ATV Dose 520mg/m^2 Capsule: Group 3 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (capsule) and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  ATV Final Recommended Dose: 520mg/m^2 Capsule
- Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV: Group 5 enrolled participants between 91 days of age and 2 years of age. They received ATV (powder), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended: 310mg/m^2
Arm/Group | Step I: Group 3: ATV Dose 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 20 | 21 | 17 | 11 | 21 | 21 | 14
ng/mL | 6463 [4994 to 8207] | 7006 [5925 to 9324] | 6501 [3218 to 9083] | 4952 [1365 to 6070] | 5593 [4151 to 7548] | 5013 [3692 to 5993] | 4095 [2947 to 5563]

9. Primary Outcome: Pharmacokinetic (PK) Parameter: Clearance (CL/F)
Description: Pharmacokinetics were determined by non-compartmental analysis and Apparent oral clearance (CL/F) was calculated as ATV dose divided by AUC0-24hr.
Time Frame: as for outcome 8
Population: Participants with intensive pharmacokinetic (PK) results at the final recommended dose for each group.
Measure: Median (Inter-Quartile Range); unit: L/hr/m^2
Groups:
- Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV: Group 6 enrolled participants between 2 years and 1 day of age and 13 years of age. They received ATV (powder), ritonavir, and two NRTIs.
  ATV: Participants received varying doses of ATV, depending on their age and weight. The medication was administered as 50 mg, 100 mg, or 200 mg capsules or a powder formulation, depending on which study arm participants were in.
  Ritonavir: Administered as 100 mg capsules or oral solution.
  ATV Final Recommended Dose: 310mg/m2
Arm/Group | Step I: Group 3: ATV Dose: 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 20 | 21 | 17 | 11 | 21 | 21 | 14
L/hr/m^2 | 12.8 [10.6 to 21.1] | 11.4 [7.5 to 14.2] | 7.9 [5.1 to 12] | 8.3 [5.6 to 22.4] | 5.3 [3.8 to 8.2] | 4.7 [3.9 to 5.9] | 4.8 [3.4 to 5.1]

10. Secondary Outcome: Change in CD4 Count (Cells/mm^3) From Baseline to Week 20
Time Frame: Baseline, Week 20
Population: Participants accrued at the final recommended dose for each group (with evaluable CD4 data).
  CD4 changes from baseline were calculated in an 'as-treated' analysis' such that only patients who tolerated the study treatment, and who had evaluable data were included in this analysis.
Measure: Median (Full Range); unit: Cells/mm^3
Arm/Group | Step I: Group 3: ATV Dose: 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 19 | 17 | 17 | 7 | 24 | 21 | 9
Cells/mm^3 | 120 [-138 to 599] | 184 [-122 to 449] | 286 [-1388 to 2306] | -294 [-858 to 1779] | 312 [-615 to 1065] | 176 [-368 to 935] | 139 [-110 to 327]

11. Secondary Outcome: Change in CD4 Count (Cells/mm^3) From Baseline to Week 48
Time Frame: Baseline, Week 48
Population: Patients accrued to the final recommended dose for each group (with evaluable CD4 data).
  CD4 changes from baseline were calculated in an 'as-treated' analysis' such that only patients who tolerated the study treatment, and who had evaluable data were included in this analysis.
Measure: Median (Full Range); unit: Cells/mm^3
Arm/Group | Step I: Group 3: ATV Dose: 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 15 | 10 | 14 | 6 | 23 | 20 | 8
Cells/mm^3 | 164 [60 to 590] | 140 [-171 to 348] | 74 [-912 to 1056] | -232 [-480 to 996] | 324 [-297 to 1833] | 157 [-306 to 1006] | 135 [-194 to 422]

12. Secondary Outcome: Change in CD4 Count (Cells/mm^3) From Baseline to Week 96
Time Frame: Baseline, Week 96
Population: as for outcome 11
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | Step I: Group 3: ATV Dose: 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 16 | 10 | 14 | 2 | 21 | 17 | 3
cells/mm^3 | 366 [-114 to 916] | 233 [92 to 410] | 340 [-938 to 1640] | -600 [-828 to -371] | 317 [28 to 1693] | 260 [-106 to 1230] | 293 [85 to 337]

13. Secondary Outcome: Change in CD4 Percent From Baseline to Week 20
Time Frame: Baseline, Week 20
Population: as for outcome 11
Measure: Median (Full Range); unit: percentage of total lymphocytes
Arm/Group | Step I: Group 3: ATV Dose: 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 19 | 17 | 17 | 7 | 24 | 22 | 9
percentage of total lymphocytes | 8 [-2 to 16] | 6 [-5 to 16] | 8 [-9 to 22] | 6 [-16 to 12] | 11 [3 to 24] | 7 [-7 to 17] | 3 [-1 to 10]

14. Secondary Outcome: Change in CD4 Percent From Baseline to Week 48
Time Frame: Baseline, Week 48
Population: as for outcome 11
Measure: Median (Full Range); unit: percentage of total lymphocytes
Arm/Group | Step I: Group 3: ATV Dose: 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 15 | 10 | 14 | 6 | 23 | 20 | 8
percentage of total lymphocytes | 7 [-3 to 18] | 9 [-1 to 15] | 10 [-4 to 20] | 0 [-14 to 12] | 12 [-1 to 30] | 8 [-6 to 26] | 5 [0 to 23]

15. Secondary Outcome: Change in CD4 Percent From Baseline to Week 96
Time Frame: Baseline, Week 96
Population: as for outcome 11
Measure: Median (Full Range); unit: percentage of total lymphocytes
Arm/Group | Step I: Group 3: ATV Dose: 520mg/m^2 Capsule | Step I: Group 4: ATV Dose: 620mg/m^2 Capsule | Step I: Group 5: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 5a: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 6: ATV Dose: 310mg/m^2 Powder + RTV | Step I: Group 7: ATV Dose: 205mg/m^2 Capsule + RTV | Step I: Group 8: ATV Dose: 205mg/m^2 Capsule + RTV
Number analyzed (Participants) | 16 | 10 | 14 | 2 | 21 | 17 | 3
percentage of total lymphocytes | 14 [1 to 26] | 9 [3 to 15] | 10 [1 to 27] | -0.5 [-1 to 0] | 15 [-1 to 32] | 10 [-10 to 35] | 9 [4 to 16]

ADVERSE EVENTS:
Time Frame: From first study enrollment (16 November 2000) up to the last off-study visit (15 September 2014)
Description: P1020A followed intensive reporting requirements defined in DAIDS Serious Adverse Experience Reporting Manual. AEs graded according to the Division of AIDS (DAIDS) AE Grading Table (see references in the Protocol Section) as follows: Gr 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Potentially Life-Threatening, Gr 5=Death.
Groups:
- Group 3: ATV 520mg/m^2 Capsule: 2 years and 1 day (731 days or more) to 13 years of age.
  ATV capsule + 2 NRTIs
  Note: This is the final recommended dose for this group.
- Group 4: ATV 620mg/m^2 Capsule: 13 years and 1 day to 21 (not including the 22nd birthday) years of age.
  ATV capsule + 2 NRTIs
  Note: This is the final recommended dose for this group.
- Group 5: ATV 310mg/m^2 Powder + RTV: 91 days to 2 years of age (less than or exactly 730 days.
  ATV powder + ritonavir + 2 NRTIs
  Note: This is the final recommended dose for this group.
- Group 6: ATV 310mg/m^2 Powder + RTV: 2 years and 1 day (731 days or more) to 13 years of age.
  ATV powder + ritonavir + 2 NRTIs
  Note: This is the final recommended dose for this group.
- Group 7: ATV 205mg/m^2 Capsule + RTV: 2 years and 1 day (731 days or more) to 13 years of age.
  ATV capsule + ritonavir + 2 NRTIs
  Note: This is the final recommended dose for this group.
- Group 8: ATV 205mg/m^2 Capsule + RTV: 13 years and 1 day to 21 (not including the 22nd birthday) years of age.
  ATV capsule + ritonavir + 2 NRTIs
  Note: This is the final recommended dose for this group.
- Group 5A: ATV 310mg/m^2 Powder + RTV: 91 to 180 days of age.
  ATV powder + ritonavir + 2 NRTIs
  Note: This is the final recommended dose for this group.
Arm/Group | Group 3: ATV 520mg/m^2 Capsule | Group 4: ATV 620mg/m^2 Capsule | Group 5: ATV 310mg/m^2 Powder + RTV | Group 6: ATV 310mg/m^2 Powder + RTV | Group 7: ATV 205mg/m^2 Capsule + RTV | Group 8: ATV 205mg/m^2 Capsule + RTV | Group 5A: ATV 310mg/m^2 Powder + RTV
Serious Adverse Events (participants affected / at risk) | 10/21 | 15/25 | 12/21 | 14/26 | 15/24 | 8/14 | 5/11
Other Adverse Events (participants affected / at risk) | 21/21 | 25/25 | 21/21 | 26/26 | 24/24 | 14/14 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 3: ATV 520mg/m^2 Capsule (N=21) | Group 4: ATV 620mg/m^2 Capsule (N=25) | Group 5: ATV 310mg/m^2 Powder + RTV (N=21) | Group 6: ATV 310mg/m^2 Powder + RTV (N=26) | Group 7: ATV 205mg/m^2 Capsule + RTV (N=24) | Group 8: ATV 205mg/m^2 Capsule + RTV (N=14) | Group 5A: ATV 310mg/m^2 Powder + RTV (N=11)
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 6 | 2 | 4 | 3 | 1 | 1
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 7 | 8 | 6 | 8 | 10 | 5 | 0
Blood bilirubin unconjugated increased (Investigations) | 1 | 6 | 5 | 8 | 9 | 2 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 0 | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial wasting (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipoatrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 3: ATV 520mg/m^2 Capsule (N=21) | Group 4: ATV 620mg/m^2 Capsule (N=25) | Group 5: ATV 310mg/m^2 Powder + RTV (N=21) | Group 6: ATV 310mg/m^2 Powder + RTV (N=26) | Group 7: ATV 205mg/m^2 Capsule + RTV (N=24) | Group 8: ATV 205mg/m^2 Capsule + RTV (N=14) | Group 5A: ATV 310mg/m^2 Powder + RTV (N=11)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2 | 1 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 7 | 10 | 11 | 7 | 7 | 1 | 6
Splenomegaly (Blood and lymphatic system disorders) | 2 | 1 | 6 | 0 | 1 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 4 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 7 | 3 | 4 | 8 | 2 | 2 | 2
Hypoacusis (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 3 | 2 | 7 | 4 | 3 | 0 | 2
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Eye discharge (Eye disorders) | 5 | 0 | 5 | 10 | 2 | 1 | 2
Eye pain (Eye disorders) | 0 | 3 | 3 | 3 | 2 | 0 | 0
Eye pruritus (Eye disorders) | 3 | 2 | 4 | 4 | 4 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 3 | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 2 | 2 | 2 | 6 | 5 | 1 | 0
Ocular icterus (Eye disorders) | 7 | 7 | 5 | 7 | 9 | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 6 | 5 | 5 | 6 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 5 | 2 | 4 | 4 | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 5 | 12 | 11 | 7 | 4 | 8
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Gingival ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 2 | 2 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 5 | 1 | 7 | 2 | 3 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 3 | 4 | 0 | 2 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal lesion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 2 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 1 | 5 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 13 | 8 | 14 | 19 | 7 | 3 | 5
Asthenia (General disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 4 | 6 | 2 | 4 | 6 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Face oedema (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 1 | 0 | 3 | 1
Pain (General disorders) | 3 | 0 | 0 | 2 | 1 | 1 | 0
Peripheral swelling (General disorders) | 2 | 3 | 1 | 1 | 5 | 1 | 0
Pyrexia (General disorders) | 14 | 8 | 15 | 16 | 9 | 6 | 8
Secretion discharge (General disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 4 | 6 | 8 | 4 | 0 | 1
Jaundice (Hepatobiliary disorders) | 2 | 3 | 2 | 1 | 2 | 1 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Serum sickness (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acarodermatitis (Infections and infestations) | 3 | 2 | 8 | 5 | 5 | 0 | 0
Acute sinusitis (Infections and infestations) | 2 | 3 | 1 | 2 | 0 | 1 | 0
Body tinea (Infections and infestations) | 1 | 0 | 6 | 3 | 2 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 6 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2 | 2 | 2 | 1 | 1 | 0
Conjunctivitis (Infections and infestations) | 6 | 0 | 4 | 6 | 5 | 0 | 2
Fungal skin infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 5 | 4 | 2 | 2 | 5
Gingivitis (Infections and infestations) | 1 | 1 | 2 | 1 | 1 | 0 | 0
Helminthic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Immune reconstitution inflammatory syndrome associated tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Impetigo (Infections and infestations) | 3 | 2 | 4 | 5 | 4 | 0 | 4
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Meningitis haemophilus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Molluscum contagiosum (Infections and infestations) | 2 | 1 | 3 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 2 | 5 | 4 | 1 | 0 | 0 | 2
Oral herpes (Infections and infestations) | 1 | 3 | 2 | 4 | 3 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 2 | 2 | 2 | 1 | 0 | 0
Otitis media (Infections and infestations) | 7 | 3 | 8 | 9 | 2 | 2 | 3
Otitis media acute (Infections and infestations) | 2 | 3 | 11 | 5 | 3 | 0 | 2
Otitis media chronic (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Parotitis (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 4 | 5 | 7 | 10 | 6 | 1 | 3
Pharyngitis streptococcal (Infections and infestations) | 4 | 0 | 1 | 2 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 3 | 8 | 6 | 7 | 0 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 2
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 2 | 0 | 0 | 1 | 1 | 0 | 2
Purulent discharge (Infections and infestations) | 2 | 0 | 2 | 2 | 1 | 0 | 4
Rash pustular (Infections and infestations) | 1 | 1 | 1 | 1 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 2
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Staphylococcal impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Streptococcal impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Tinea capitis (Infections and infestations) | 3 | 0 | 8 | 6 | 2 | 0 | 1
Tinea faciei (Infections and infestations) | 2 | 0 | 3 | 1 | 3 | 0 | 0
Tinea infection (Infections and infestations) | 9 | 0 | 7 | 3 | 3 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinea versicolour (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 5 | 4 | 8 | 9 | 4 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 1 | 1 | 2 | 3 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 13 | 14 | 14 | 15 | 15 | 5 | 7
Aspartate aminotransferase increased (Investigations) | 12 | 16 | 14 | 15 | 19 | 5 | 5
Bilirubin conjugated increased (Investigations) | 14 | 13 | 13 | 19 | 19 | 7 | 5
Blood alkaline phosphatase increased (Investigations) | 7 | 5 | 4 | 6 | 8 | 1 | 0
Blood bilirubin (Investigations) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 12 | 12 | 12 | 18 | 13 | 7 | 8
Blood bilirubin unconjugated (Investigations) | 1 | 1 | 1 | 3 | 1 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 19 | 16 | 14 | 18 | 14 | 11 | 8
Blood calcium abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Blood calcium decreased (Investigations) | 0 | 2 | 0 | 1 | 1 | 0 | 0
Blood calcium increased (Investigations) | 0 | 2 | 3 | 3 | 0 | 1 | 2
Blood cholesterol abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood cholesterol increased (Investigations) | 10 | 11 | 17 | 22 | 13 | 7 | 7
Blood creatine phosphokinase increased (Investigations) | 6 | 1 | 3 | 1 | 2 | 1 | 2
Blood creatinine increased (Investigations) | 13 | 5 | 6 | 8 | 11 | 4 | 3
Blood glucose abnormal (Investigations) | 2 | 2 | 3 | 3 | 4 | 1 | 1
Blood glucose decreased (Investigations) | 15 | 18 | 16 | 22 | 14 | 3 | 6
Blood glucose increased (Investigations) | 7 | 9 | 4 | 10 | 8 | 3 | 2
Blood magnesium decreased (Investigations) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Blood potassium abnormal (Investigations) | 6 | 6 | 14 | 12 | 12 | 1 | 9
Blood potassium decreased (Investigations) | 10 | 7 | 10 | 13 | 8 | 4 | 3
Blood potassium increased (Investigations) | 6 | 9 | 17 | 18 | 9 | 1 | 7
Blood sodium abnormal (Investigations) | 1 | 3 | 1 | 0 | 1 | 1 | 1
Blood sodium decreased (Investigations) | 17 | 17 | 17 | 23 | 18 | 5 | 10
Blood sodium increased (Investigations) | 4 | 4 | 3 | 2 | 6 | 1 | 1
Blood triglycerides increased (Investigations) | 19 | 19 | 20 | 25 | 19 | 7 | 10
Blood urea abnormal (Investigations) | 4 | 4 | 2 | 4 | 3 | 0 | 4
Blood uric acid increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Breath sounds abnormal (Investigations) | 3 | 1 | 3 | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 6 | 12 | 12 | 14 | 10 | 5 | 5
Haemoglobin decreased (Investigations) | 11 | 11 | 14 | 21 | 12 | 3 | 6
High density lipoprotein abnormal (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Low density lipoprotein abnormal (Investigations) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 11 | 11 | 19 | 17 | 14 | 7 | 8
Pancreatic enzymes abnormal (Investigations) | 0 | 2 | 7 | 1 | 3 | 1 | 0
Weight decreased (Investigations) | 3 | 4 | 3 | 2 | 5 | 0 | 1
Abnormal weight gain (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | 7 | 10 | 4 | 1 | 5
Failure to thrive (Metabolism and nutrition disorders) | 1 | 3 | 3 | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 2 | 1 | 1 | 1
Clubbing (Musculoskeletal and connective tissue disorders) | 4 | 1 | 4 | 6 | 3 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4 | 3 | 3 | 4 | 2 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 2 | 2 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 4 | 0 | 0 | 1 | 1 | 1
Epilepsy (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 9 | 7 | 3 | 6 | 4 | 2 | 1
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Agoraphobia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anger (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 3 | 1 | 3 | 0 | 0
Depression (Psychiatric disorders) | 1 | 2 | 0 | 1 | 0 | 3 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Panic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 2 | 0 | 0
Enuresis (Renal and urinary disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Perineal rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 3 | 0 | 3 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Vulval disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 | 1 | 0 | 1 | 3 | 0 | 0
Vulvovaginal rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 5 | 2 | 0 | 0 | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 5 | 2 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 16 | 19 | 26 | 18 | 9 | 9
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 7 | 2 | 0 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4 | 2 | 2 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 10 | 14 | 7 | 3 | 4
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 5 | 11 | 7 | 3 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 3 | 5 | 1 | 1 | 2
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 5 | 6 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 13 | 7 | 13 | 19 | 7 | 4 | 7
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 | 1 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3 | 1 | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 4 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4 | 8 | 4 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 3 | 1 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 1 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 1 | 0 | 0 | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 0 | 2 | 4 | 3 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 3 | 4 | 7 | 6 | 4 | 0 | 3
Eosinophilic pustular folliculitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 0 | 3 | 1 | 0 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial wasting (Skin and subcutaneous tissue disorders) | 1 | 0 | 6 | 5 | 3 | 0 | 0
Lipoatrophy (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 1 | 1 | 0
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 1
Pityriasis alba (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 3 | 3 | 2 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 12 | 11 | 16 | 13 | 11 | 4 | 7
Rash generalised (Skin and subcutaneous tissue disorders) | 3 | 3 | 7 | 7 | 3 | 1 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 3 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 7 | 0 | 8 | 12 | 9 | 0 | 3
Skin plaque (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 4 | 0 | 0
Umbilical haematoma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.